CLINICAL TRIAL: NCT06000826
Title: Efficacy of a Low-cost Warming Mattress Celsi Warmer for the Management of Hypothermic Newborns
Brief Title: Efficacy of Celsi Warmer for the Management of Hypothermic Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: William Marsh Rice University (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-271
Record Dates: First submitted 2023-05-31; First posted 2023-08-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Newborn Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neonatal (Experimental): * A trained study nurse or clinician will transfer the enrolled participant to the study location and place the infant on the Celsi Warmer mattress.
  * A trained study nurse or clinician will attach the Celsi Warmer temperature sensor to the abdomen and secure it with the abdominal belt according to the device's instruction manual
  * A trained study nurse or clinician will wrap the baby according to the standard care at the hospital.
  * Study personnel may observe the participant during the intervention period and annotate timestamped events that might affect temperature measurement and/or thermoregulation support intervention.
  * Study personnel will perform routine abdominal skin assessments as often as every two hours and at least every 8 hours to observe for skin irritation or indentation.
  * Thermoregulation support intervention will be provided as long as the infant continues to meet criteria for continued care at clinician's discretion.
  Interventions: Device: Celsi Warmer

INTERVENTIONS:
Device: Celsi Warmer — During the study, research participants will receive thermal care via the Celsi Warmer. Aside from thermal treatment, research participants will receive the standard of care from the neonatal unit, and will also be closely monitored by study personnel throughout the study. The results from this study will allow the research team to determine if the Celsi Warmer is an effective tool for warming and monitoring newborns in wards of low-resource hospitals. The research team hopes to demonstrate that the Celsi Warmer is effective for the appropriate treatment of newborn hypothermia in hospitals in low-resource settings.

SUMMARY:
The purpose of the study is to evaluate the efficacy of a novel low-cost warming device to provide thermal care for newborn babies with hypothermia in low-resource hospitals. During the study, research participants will receive thermal care via the Celsi Warmer. Aside from thermal treatment, research participants will receive the standard of care from the neonatal unit, and will also be closely monitored by study personnel throughout the study. The results from this study will allow us to determine if the Celsi Warmer is an effective tool for warming and monitoring newborns in wards of low-resource hospitals. The research team hopes to demonstrate that the Celsi Warmer is effective for the appropriate treatment of newborn hypothermia in hospitals in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Is currently being treated at study location
* Is an inborn admission to the neonatal ward
* Whose parents or guardians provided a written informed consent
* Whose parents or guardians providing informed consent are 18 years old or older
* Has a current weight of greater than or equal to 1.0 kg and less than or equal to 4.0kg
* Has been identified as in need of thermal care defined as having a moderate hypothermic temperature (32.0-36.0°C) as the last temperature recorded in hospital chart, or during recruitment procedures; and
* Is unable to be enrolled in KMC for reasons including, but not limited to:

  1. Mother/guardian unable or unavailable to provide KMC
  2. Under observation in NICU before transfer to KMC
  3. No space in KMC
  4. Clinician's discretion
* May be receiving other medical treatments, including but not limited to, CPAP, oxygen therapy, IV fluids, management and monitoring of common newborn conditions such as hypoglycemia, and/or hyperbilirubinemia via LED phototherapy

Exclusion Criteria:

* Requires mechanical ventilation
* deemed in need of intensive care by the hospital staff who is providing care,including but not limited to:

  1. Neonates with severe anemia and/or any suspected hematological disorders, and/or
  2. Neonates with obvious congenital anomalies, and/or
  3. neonates suspected with hypo/hyperthyroidism or any hormonal disorders
* Has been diagnosed with birth asphyxia
* Presents a condition that precludes the use of the temperature sensor and/or abdominal belt including but not limited to, gastroschisis, known umbilical cord infection, known skin infection
* Whose clinician presents concerns about their participation
* Is receiving treatment that participation in the study would interfere with, i.e.transferring to KMC

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Broad Objective - Comparison to the Gold Standard of Rewarming Hypothermic Newborns | 1 year
  To evaluate the clinical efficacy and safety of the Celsi Warmer in rewarming hypothermic newborns by comparing the Celsi Warmer's accuracy in measuring neonatal temperature compared to the gold standard, axillary temperature readings.

SECONDARY OUTCOMES:
Efficacy of the Device | 1 year
  To assess the performance of the Celsi Warmer in rewarming hypothermic newborns by measuring the incidence of attainment of normothermia (36.5-37.5°C)
Safety of the Device - Measure of Infant's Increase in Temperature | 1 year
  To measure the infant's rate of temperature (°C) increase through thermoregulatory intervention.
Safety of the Device - Local Effect of the Abdominal Belt | 1 year
  To evaluate the local effect of the abdominal belt on newborn's skin by looking at any evidence of skin irritation
Safety of the Device - Incidence of Hyperthermia | 1 year
  To evaluate any incidence of hyperthermia (>37.5°C) during the thermoregulation intervention.
Safety of the Device - Incidence of Rebound Hypothermia | 1 year
  To report any incidence of rebound hypothermia ( < 36.5°C) (post-intervention hypothermia) up to 72 hours from the initial encounter.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R Richards-Kortum, PhD, Principal Investigator — William Marsh Rice University
Locations (1):
- Muhimbili University of Health and Allied Sciences (MUHAS), Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar V, Shearer JC, Kumar A, Darmstadt GL. Neonatal hypothermia in low resource settings: a review. J Perinatol. 2009 Jun;29(6):401-12. doi: 10.1038/jp.2008.233. Epub 2009 Jan 22. PMID 19158799
- [Background] Carns J, Kawaza K, Quinn MK, Miao Y, Guerra R, Molyneux E, Oden M, Richards-Kortum R. Impact of hypothermia on implementation of CPAP for neonatal respiratory distress syndrome in a low-resource setting. PLoS One. 2018 Mar 15;13(3):e0194144. doi: 10.1371/journal.pone.0194144. eCollection 2018. PMID 29543861
- [Background] Cavallin F, Calgaro S, Brugnolaro V, Seni AHA, Muhelo AR, Da Dalt L, Putoto G, Trevisanuto D. Impact of temperature change from admission to day one on neonatal mortality in a low-resource setting. BMC Pregnancy Childbirth. 2020 Oct 23;20(1):646. doi: 10.1186/s12884-020-03343-7. PMID 33097025
- [Background] Mullany LC. Neonatal hypothermia in low-resource settings. Semin Perinatol. 2010 Dec;34(6):426-33. doi: 10.1053/j.semperi.2010.09.007. PMID 21094417
- [Background] Lunze K, Bloom DE, Jamison DT, Hamer DH. The global burden of neonatal hypothermia: systematic review of a major challenge for newborn survival. BMC Med. 2013 Jan 31;11:24. doi: 10.1186/1741-7015-11-24. PMID 23369256
- [Background] Manji KP, Kisenge R. Neonatal hypothermia on admission to a special care unit in Dar-es-Salaam, Tanzania: a cause for concern. Cent Afr J Med. 2003 Mar-Apr;49(3-4):23-7. PMID 14562586
- [Background] Laptook AR, Salhab W, Bhaskar B; Neonatal Research Network. Admission temperature of low birth weight infants: predictors and associated morbidities. Pediatrics. 2007 Mar;119(3):e643-9. doi: 10.1542/peds.2006-0943. Epub 2007 Feb 12. PMID 17296783
- [Background] Lunze K, Hamer DH. Thermal protection of the newborn in resource-limited environments. J Perinatol. 2012 May;32(5):317-24. doi: 10.1038/jp.2012.11. Epub 2012 Mar 1. PMID 22382859
- [Background] de Almeida MF, Guinsburg R, Sancho GA, Rosa IR, Lamy ZC, Martinez FE, da Silva RP, Ferrari LS, de Souza Rugolo LM, Abdallah VO, Silveira Rde C; Brazilian Network on Neonatal Research. Hypothermia and early neonatal mortality in preterm infants. J Pediatr. 2014 Feb;164(2):271-5.e1. doi: 10.1016/j.jpeds.2013.09.049. Epub 2013 Nov 6. PMID 24210925
- [Background] ADAMSON SK Jr, TOWELL ME. THERMAL HOMEOSTASIS IN THE FETUS AND NEWBORN. Anesthesiology. 1965 Jul-Aug;26:531-48. doi: 10.1097/00000542-196507000-00017. No abstract available. PMID 14313463
- [Background] Nahimana E, May L, Gadgil A, Rapp V, Magge H, Kubwimana M, Nshimyiryo A, Kateera F, Feldman HA, Nkikabahizi F, Sayinzoga F, Hansen A. A low cost, re-usable electricity-free infant warmer: evaluation of safety, effectiveness and feasibiliy. Public Health Action. 2018 Dec 21;8(4):211-217. doi: 10.5588/pha.18.0031. PMID 30775282
- [Background] Wyllie J, Perlman JM, Kattwinkel J, Wyckoff MH, Aziz K, Guinsburg R, Kim HS, Liley HG, Mildenhall L, Simon WM, Szyld E, Tamura M, Velaphi S; Neonatal Resuscitation Chapter Collaborators. Part 7: Neonatal resuscitation: 2015 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Resuscitation. 2015 Oct;95:e169-201. doi: 10.1016/j.resuscitation.2015.07.045. Epub 2015 Oct 15. No abstract available. PMID 26477424
- [Background] Wyckoff MH, Wyllie J, Aziz K, de Almeida MF, Fabres J, Fawke J, Guinsburg R, Hosono S, Isayama T, Kapadia VS, Kim HS, Liley HG, McKinlay CJD, Mildenhall L, Perlman JM, Rabi Y, Roehr CC, Schmolzer GM, Szyld E, Trevisanuto D, Velaphi S, Weiner GM; Neonatal Life Support Collaborators. Neonatal Life Support: 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2020 Oct 20;142(16_suppl_1):S185-S221. doi: 10.1161/CIR.0000000000000895. Epub 2020 Oct 21. PMID 33084392
- [Background] WHO Immediate KMC Study Group; Arya S, Naburi H, Kawaza K, Newton S, Anyabolu CH, Bergman N, Rao SPN, Mittal P, Assenga E, Gadama L, Larsen-Reindorf R, Kuti O, Linner A, Yoshida S, Chopra N, Ngarina M, Msusa AT, Boakye-Yiadom A, Kuti BP, Morgan B, Minckas N, Suri J, Moshiro R, Samuel V, Wireko-Brobby N, Rettedal S, Jaiswal HV, Sankar MJ, Nyanor I, Tiwary H, Anand P, Manu AA, Nagpal K, Ansong D, Saini I, Aggarwal KC, Wadhwa N, Bahl R, Westrup B, Adejuyigbe EA, Plange-Rhule G, Dube Q, Chellani H, Massawe A. Immediate "Kangaroo Mother Care" and Survival of Infants with Low Birth Weight. N Engl J Med. 2021 May 27;384(21):2028-2038. doi: 10.1056/NEJMoa2026486. PMID 34038632
- [Background] Ahmed S, Mitra SN, Chowdhury AM, Camacho LL, Winikoff B, Sloan NL. Community Kangaroo Mother Care: implementation and potential for neonatal survival and health in very low-income settings. J Perinatol. 2011 May;31(5):361-7. doi: 10.1038/jp.2010.131. Epub 2011 Feb 10. PMID 21311502
- [Background] Lee HC, Martin-Anderson S, Dudley RA. Clinician perspectives on barriers to and opportunities for skin-to-skin contact for premature infants in neonatal intensive care units. Breastfeed Med. 2012 Apr;7(2):79-84. doi: 10.1089/bfm.2011.0004. Epub 2011 Oct 19. PMID 22011130
- [Background] Flenady VJ, Woodgate PG. Radiant warmers versus incubators for regulating body temperature in newborn infants. Cochrane Database Syst Rev. 2000;2003(2):CD000435. doi: 10.1002/14651858.CD000435. PMID 10796363
- [Background] Trevisanuto D, Coretti I, Doglioni N, Udilano A, Cavallin F, Zanardo V. Effective temperature under radiant infant warmer: does the device make a difference? Resuscitation. 2011 Jun;82(6):720-3. doi: 10.1016/j.resuscitation.2011.02.019. Epub 2011 Mar 24. PMID 21439704
- [Background] Butin M, Dumont Y, Monteix A, Raphard A, Roques C, Martins Simoes P, Picaud JC, Laurent F. Sources and reservoirs of Staphylococcus capitis NRCS-A inside a NICU. Antimicrob Resist Infect Control. 2019 Oct 17;8:157. doi: 10.1186/s13756-019-0616-1. eCollection 2019. PMID 31636900
- [Background] Cadot L, Bruguiere H, Jumas-Bilak E, Didelot MN, Masnou A, de Barry G, Cambonie G, Parer S, Romano-Bertrand S. Extended spectrum beta-lactamase-producing Klebsiella pneumoniae outbreak reveals incubators as pathogen reservoir in neonatal care center. Eur J Pediatr. 2019 Apr;178(4):505-513. doi: 10.1007/s00431-019-03323-w. Epub 2019 Jan 23. PMID 30671695
- [Background] Nimbalkar S, Patel H, Dongara A, Patel DV, Bansal S. Usage of EMBRACE(TM) in Gujarat, India: Survey of Paediatricians. Adv Prev Med. 2014;2014:415301. doi: 10.1155/2014/415301. Epub 2014 Oct 30. PMID 25530887
- [Background] Boo NY, Selvarani S. Effectiveness of a simple heated water-filled mattress for the prevention and treatment of neonatal hypothermia in the labour room. Singapore Med J. 2005 Aug;46(8):387-91. PMID 16049607
- [Background] McNichol L, Lund C, Rosen T, Gray M. Medical adhesives and patient safety: state of the science: consensus statements for the assessment, prevention, and treatment of adhesive-related skin injuries. J Wound Ostomy Continence Nurs. 2013 Jul-Aug;40(4):365-80; quiz E1-2. doi: 10.1097/WON.0b013e3182995516. PMID 23759927
- [Background] Uwamariya J, Mazimpaka C, May L, Nshimyiryo A, Feldman HA, Sayinzoga F, Umutesi S, Gadgil A, Rapp VH, Nahimana E, Hansen A. Safety and effectiveness of a non-electric infant warmer for hypothermia in Rwanda: A cluster-randomized stepped-wedge trial. EClinicalMedicine. 2021 Apr 16;34:100842. doi: 10.1016/j.eclinm.2021.100842. eCollection 2021 Apr. PMID 33997734